CLINICAL TRIAL: NCT00922805
Title: Soluble Fiber Use in Pediatric Short Bowel Syndrome
Brief Title: Fiber Use in Pediatric Short Bowel Syndrome
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Collaborators: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency); Baylor College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CUMG-108061
Record Dates: First submitted 2009-06-16; First posted 2009-06-17 (Estimated); Last update posted 2014-01-15 (Estimated); Status verified 2014-01

CONDITIONS: Short Bowel Syndrome
Keywords: Pediatrics, short bowel syndrome, soluble fiber
MeSH Terms: conditions — Short Bowel Syndrome | interventions — guar gum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- fiber-enriched formula then fiber-free formula (Active Comparator): Subjects first receive a fiber-enriched formula for one week but then will be crossed over and receive a fiber-free formula
  Interventions: Dietary Supplement: guar gum
- fiber-free formula then fiber-enriched formula (Active Comparator): Subjects receive first formula only then will be crossed over and receive a fiber-enriched formula
  Interventions: Dietary Supplement: guar gum

INTERVENTIONS:
Dietary Supplement: guar gum — guar gum (20 g/l of formula) for one week
  Other Names: Benefiber

SUMMARY:
Short bowel syndrome (SBS) is a form of disease that results from removal of a significant portion of the intestine leading to poor nutrient absorption. Infants with short bowel syndrome suffer from diarrhea and poor growth. The care of these infants is limited by the lack of effective therapies.

Soluble fiber (guar gum) is an indigestible form of sugar that is mostly contained in fruits and vegetables. Soluble fiber can reduce the severity and duration of persistent (constant) diarrhea in children.

The purpose of this research study is to evaluate the many effects of fiber added in the diet of infants with SBS

DETAILED DESCRIPTION:
Short bowel syndrome (SBS) is a form of disease that results from removal of a significant portion of the intestine leading to poor nutrient absorption. Infants with short bowel syndrome suffer from diarrhea and poor growth. The care of these infants is limited by the lack of effective therapies. As the intestine tries to grow back some of its length, a process that can take many months, these infants become dependent on intravenous (IV) nutrition in order to survive. Liver disease and sepsis (a blood stream infection) are common complications of IV nutrition and are the two most common causes of death in this population. Therefore, clinicians have tried different ways to improve feeding and shorten the amount of time of IV nutrition, for example continuous feedings through the intestine, use of partly digested formulas and change in diet.

Soluble fiber (guar gum) is an indigestible form of sugar that is mostly contained in fruits and vegetables. Soluble fiber can reduce the severity and duration of persistent (constant) diarrhea in children.

The purpose of this research study is to evaluate the many effects of fiber added in the diet of infants with SBS.

ELIGIBILITY:
Pediatric infants (less than 1 y of age) who

1. Have Short Bowel Syndrome defined by a history of congenital or surgical loss of intestinal absorptive function resulting in parenteral nutrition dependency of longer than 30 days;
2. Are receiving at least 20% of their caloric needs from enteral nutrition and have been on enteral nutrition for at least 1 week following intestinal resection;
3. Have increased stool output as manifested by watery stools (3-12/day) and increased ostomy output (20-50 cc/kg/day);
4. Have not received antibiotics, probiotics or prebiotics for 2 weeks prior to study entry;

Ages: 2 Weeks to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2009-01; Primary Completion 2012-01 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Soluble fiber supplementation, as a short chain fatty acid precursor, will improve intestinal integrity of infants with SBS | 4 weeks

SECONDARY OUTCOMES:
Soluble fiber supplementation will improve enteral energy intake of infants with SBS | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Juliana C Frem, MD, Principal Investigator — University of Arkansas
Locations (1):
- Arkansas Children's Hospital, Little Rock, Arkansas, United States